CLINICAL TRIAL: NCT02208180
Title: Heart Healthy Lenoir: Return of Results Study
Acronym: HHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Harlyn Skinner, MS, Doctoral Candidate, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-1500; 1P50HL105184-01 (NIH)
Record Dates: First submitted 2014-07-30; First posted 2014-08-04 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Disease
Keywords: Return of results; Genomics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Return of genomic results on cardiovascular disease risk (Experimental): Participants will receive genomic cardiovascular disease risk information.
  Interventions: Behavioral: Return of genomic results on cardiovascular disease risk
- Return of lifestyle results on cardiovascular disease risk (Active Comparator): Participants will receive lifestyle cardiovascular disease risk information. Genomic risk information will be returned after the conclusion of the study.
  Interventions: Behavioral: Return of genomic results on cardiovascular disease risk

INTERVENTIONS:
Behavioral: Return of genomic results on cardiovascular disease risk — Experimental group: Participants will receive genomic cardiovascular disease risk information.
  Comparator: Participants will receive lifestyle cardiovascular disease risk information. Genomic risk information will be returned after the conclusion of the study.

SUMMARY:
The investigators are conducting a two group intervention to study to the effect of individualized heart disease genomic risk results on motivation towards diet and physical activity behaviors to reduce heart disease risk. The intervention includes provided participants with genomic and lifestyle risk estimates. Investigators will follow participants for 3 months to determine if motivation towards and engagement in diet and physical activity behaviors change.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Heart Healthy Lenoir Genomics
* African-American (self-identified)
* Wants to be contacted for future studies

Exclusion Criteria:

* Enrolled in an arm of the Heart Healthy Lenoir Lifestyle study with intense behavioral intervention (e.g. weight loss or weight maintenance programs)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in motivation | Baseline, Post-interview, 3 months
  The Prevention and Planning Behaviors Scale is a recently developed tool that provides a direct measure of degrees of influence on participants' motivation to change their health behavior in translational genomic studies. It has 23-items where participants rate themselves using a 5-point Likert scale (1=A Lot Less Motivated to 5=A Lot More Motivated).

SECONDARY OUTCOMES:
Change in Eating Habits | Baseline, 3 months
  Eating habits will be assessed using a 10-item Block questionnaire designed to capture the frequency with which participants eat particular items from different food groups. Participants will rate themselves on a 6-point scale ranging from "Less than 1 time per WEEK" to "2+ a DAY."
Change in Physical Activity | Baseline, 3 months
  The 16-item RESIDE Neighborhood Physical Activity Questionnaire will be used to assess context-specific walking behavior through self-report. Participants are asked how often they walk, how long, to where, and similar questions about what other types of physical activity they might engage in. Giles-Corti B, Timperio A, Cutt H, Pikora TJ, Bull FC, Knuiman M, et al. Development of a reliable measure of walking within and outside the local neighborhood: RESIDE's Neighborhood Physical Activity Questionnaire. Preventive medicine 2006;42(6):455-459.

OTHER OUTCOMES:
Change in Psychological Adaptation | Baseline, 3 months
  The Psychological Adaptation Scale (PAS) measures adaptation to health risk information via a 20-item questionnaire rated on a 5-point Likert scale (1=Not At All to 5=Very Much). This questionnaire measures adaptation in 4 domains: coping efficacy, self-esteem, social integration, and spiritual well-being. This scale was developed specifically for use in genomic studies to measure adaptation and aid understanding in the relationship between health outcomes and psychological well-being. Biesecker BB, Erby LH, Woolford S, Adcock JY, Cohen JS, Lamb A, et al. Development and validation of the Psychological Adaptation Scale (PAS): Use in six studies of adaptation to a health condition or risk. Patient Educ Couns 2013.

CONTACTS AND LOCATIONS:
Overall Officials: Harlyn G Skinner, MS, Principal Investigator — University of North Carolina, Chapel Hill; Alice Ammerman, DrPH, MPH, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- Heart Healthy Lenoir Field Office, Kinston, North Carolina, United States